CLINICAL TRIAL: NCT02052908
Title: A Phase Ib Biomarker Trial of Naproxen in Patients at Risk for DNA Mismatch Repair Deficient Colorectal Cancer
Brief Title: Naproxen in Preventing DNA Mismatch Repair Deficient Colorectal Cancer in Patients With Lynch Syndrome
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NCI-2014-00046; NCI-2014-00046 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); N01-CN-2012-00034; HHSN261201200034I; HUM00079757; HHSN26100003; RFP B; MDACC IRB # 2013-0698; 2013-0698; 13-585; 2013-0698 (Other: M D Anderson Cancer Center); MDA2013-01-02 (Other: DCP); N01CN00034 (NIH); P30CA016672 (NIH); NCT02048735 (obsolete NCT alias)
Record Dates: First submitted 2014-01-30; First posted 2014-02-03 (Estimated); Last update posted 2021-01-25 (Actual); Status verified 2021-01

CONDITIONS: Lynch Syndrome
MeSH Terms: conditions — Colorectal Neoplasms, Hereditary Nonpolyposis | interventions — Naproxen

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm I (high-dose naproxen) (Experimental): Patients receive high-dose naproxen PO QD for 6 months.
  Interventions: Other: Laboratory Biomarker Analysis; Drug: Naproxen
- Arm II (low-dose naproxen, placebo) (Experimental): Patients receive low-dose naproxen PO QD and placebo PO QD for 6 months.
  Interventions: Other: Laboratory Biomarker Analysis; Drug: Naproxen; Other: Placebo Administration
- Arm III (placebo) (Placebo Comparator): Patients receive placebo PO QD for 6 months.
  Interventions: Other: Laboratory Biomarker Analysis; Other: Placebo Administration

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Naproxen — Given PO
  Other Names: Naprosyn; RS-3540
  Arms: Arm I (high-dose naproxen); Arm II (low-dose naproxen, placebo)
Other: Placebo Administration — Given PO
  Arms: Arm II (low-dose naproxen, placebo); Arm III (placebo)

SUMMARY:
This randomized phase Ib trial studies the side effects and best dose of naproxen in preventing deoxyribonucleic acid (DNA) mismatch repair deficient colorectal cancer in patients with Lynch syndrome. Chemoprevention is the use of certain drugs to keep cancer from forming. The use of naproxen may keep cancer from forming in patients with Lynch syndrome.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine whether treatment with naproxen at a once-daily 220 mg or 440-mg dose, administered for 6 months as compared to placebo reduces the concentration of prostaglandin E2 (PGE2) levels in normal colorectal mucosa in subjects at risk for a mismatch repair deficient colorectal cancer.

II. To determine the toxicity profile and tolerability of naproxen at two doses (220 mg or 440-mg once daily) as compared to placebo over 6 months of therapy in subjects at risk for a mismatch repair deficient colorectal cancer.

SECONDARY OBJECTIVES:

I. To determine naproxen concentrations in plasma of patients at risk for DNA mismatch repair deficient colorectal cancer taking naproxen once daily, 220 mg, 440 mg or placebo after 6 months of therapy compared to baseline levels.

II. To determine naproxen concentrations in normal colorectal mucosa of patients at risk for DNA mismatch repair deficient colorectal cancers (CRC) taking naproxen once daily 220 mg, 440 mg or placebo after 6 months of therapy compared to baseline levels.

III. To determine whether urinary prostaglandin-endoperoxide synthase 1 metabolite (PGE-M) is significantly higher in patients at risk for DNA mismatch repair deficient CRC taking naproxen one daily, 220 mg, 440 mg or placebo after 6 months of therapy compared to baseline levels.

IV. To determine whether 6-months therapy with naproxen once daily, 220 mg, 440 mg or placebo leads to a reduction in the number of polyps observed in the rectosigmoid and rectal area.

V. To determine whether naproxen once daily, 220 mg, 440 mg or placebo will significantly change the micro-ribonucleic (RNA) profile of normal colorectal mucosa in patients at risk for DNA mismatch repair deficient CRC compared to the baseline.

VI. To determine whether naproxen once daily, 220 mg, 440 mg or placebo will significantly change the gene expression messenger RNA (mRNA) profile of normal colorectal mucosa in patients at risk for DNA mismatch repair deficient CRC compared to the baseline.

VII. To determine whether naproxen once daily, 220 mg, 440 mg or placebo will significantly change the mutational rate in patients at risk for DNA mismatch repair deficient CRC compared to placebo.

VIII. To determine future candidate biomarkers measured by genomic and transcriptomic platforms in tissue biopsies of normal colorectal mucosa in individuals at risk for mismatch repair deficient CRC pre- and post-treatment with naproxen.

IX. To determine whether Naproxen once daily, 220 mg, 440 mg or placebo will significantly change the microbiome profile of normal colorectal mucosa in patients at risk for DNA mismatch repair deficient CRC compared to the baseline.

X. To determine whether treatment with Naproxen once daily, 220 mg, 440 mg after 6 months of therapy as compared to placebo changed PGF2, PGD2, Thromboxane B2, 9a11b-PGF2a and 6-KetoPGF1a levels in colorectal mucosa of subjects at risk for a mismatch repair deficient colorectal cancer.

XI. To determine whether treatment with Naproxen once daily, 220 mg, 440 mg after 6 months of therapy as compared to placebo changed the number of stem cells and induced differentiation into other cell lineages in colorectal mucosa of subjects at risk for mismatch repair deficient colorectal cancer.

XII. To determine whether treatment with naproxen once daily, 220 mg, 440 mg after 6 months of therapy as compared to placebo changed the number of immune and mesenchymal cells recruited to the colorectal mucosa of subjects at risk for mismatch repair deficient colorectal cancer.

OUTLINE: Patients are randomized to 1 of 3 treatment arms.

ARM I: Patients receive high-dose naproxen orally (PO) once daily (QD) for 6 months.

ARM II: Patients receive low-dose naproxen PO QD and placebo PO QD for 6 months.

ARM III: Patients receive placebo PO QD for 6 months.

After completion of study treatment, patients are followed up for 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have Lynch syndrome defined as meeting any of the following:

  * "Mutation-positive Lynch syndrome": carriers or obligate carriers (by pedigree) of a pathogenic mutation in one of the DNA mismatch repair (MMR) genes (i.e. mutL homolog 1 [MLH1], mutS homolog 2 [MSH2]/epithelial cell adhesion molecule [EPCAM], mutS homolog 6 [MSH6], or PMS2 postmeiotic segregation increased 2 [S. cerevisiae] [PMS2]) or
  * "Mutation-negative Lynch syndrome": patients with a personal history of a non-sporadic MMR deficient premalignant lesion (i.e. polyp) or a non-sporadic MMR deficient malignant tumor (where "non-sporadic MMR deficient" is defined by: microsatellite-instability high by either immunohistochemistry or microsatellite instability [MSI] testing or both, but no evidence of MLH1 promoter methylation in cases with loss of both MLH1 and PMS2, and/or no evidence of v-raf murine sarcoma viral oncogene homolog B [BRAF] mutation in cases with loss of both MLH1 and PMS2) but germline MMR genetic testing showed either a variant of unknown significance or mutation negative result or had declined germline MMR genetic testing
* Participants must not have evidence of active/recurrent malignant disease for 6 months
* Participants must be at least 6 months from any prior cancer-directed treatment (such as surgical resection, chemotherapy, immunotherapy, hormonal therapy or radiation)
* Participants must have endoscopically accessible distal colon and/or rectal mucosa (i.e. participants must have at least part of the descending/sigmoid colon and/or rectum intact)
* Participants must consent to one standard of care lower gastrointestinal (GI) endoscopy (flexible sigmoidoscopy or colonoscopy) with biopsies and one flexible sigmoidoscopy with biopsies that will be 6 months (+14 days) apart
* Participants must consent to refrain from using aspirin or non-steroidal anti-inflammatory drugs (NSAIDs) or cyclooxygenase (COX)-inhibitors for the duration of the trial
* Eastern Cooperative Oncology Group (ECOG) performance status =< 1 (Karnofsky >= 70%)
* Hemoglobin >= 10 g/dL or hematocrit >= 30%
* Leukocyte count >= 3,000/microliter
* Platelet count >= 100,000/microliter
* Absolute neutrophil count >= 1,500/microliter
* Creatinine =< 1.5 x institutional upper limit of normal (ULN) (OR glomerular filtration rate [GFR] > 30 ml/min/1.73 m^2)
* Total bilirubin =< 2 x institutional ULN
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) =< 2.5 x institutional ULN
* Alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x institutional ULN
* The effects of naproxen on the developing human fetus at the recommended therapeutic dose are unknown; for this reason and because NSAIDs are known to be teratogenic, women of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) for the duration of study participation; should a woman become pregnant or suspect she is pregnant at the time of study entry or while participating in this study, she should inform her study physician immediately; women of childbearing potential must agree to baseline and pre-drug pregnancy tests
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Individuals who received scheduled aspirin, NSAIDs, or COX-inhibitors of any kind for more than 3 days (> 3 days) during anytime within the 2 weeks preceding baseline eligibility screening visit; individuals on cardio-protective aspirin will not be eligible
* Individuals who are status post total proctocolectomy (i.e. removal of all colon and rectum)
* Individuals with active gastroduodenal ulcer disease in the preceding 5 years
* Individuals with any history of transfusion-dependent gastrointestinal bleeding, gastrointestinal perforation or gastrointestinal obstruction; if any of these events had been due to a malignancy of the GI tract and the malignancy has since been removed, the patient is eligible
* Individuals with history of myocardial infarction, stroke, coronary-artery bypass draft, invasive coronary revascularization in the preceding 5 years
* Individuals taking the drugs listed below may not be randomized unless they are willing to stop the medications (and possibly change to alternative non-excluded medications to treat the same conditions) no less than 7 days prior to starting naproxen or placebo on this study; consultation with the participant's primary care provider may be obtained but is not required; the use of the following drugs or drug classes is prohibited during naproxen/placebo treatment:

  * Investigational agents
  * NSAIDs: such as aspirin, ketorolac and others NSAIDs
  * COX-2 inhibitors: such as celecoxib, rofecoxib and other COX-2
  * Antiplatelet agents: such as aspirin, clopidogrel, ticlopidine, dipyridamole, abciximab, tirofiban, eptifibatide and prasugrel
  * Anticoagulants:

    * Heparin
    * Heparinoids: such as fondaparinux, danaparoid and other heparinoids
    * Low-molecular weight heparins: such as enoxaparin, dalteparin, parnaparin, reviparin, tinzaparin, ardeparin, certoparin, lepirudin, bivalirudin
    * Other anticoagulants: argatroban, apixaban, dabigatran, rivaroxaban, warfarin, acenocoumarol, dicumarol, phenindione and other anticoagulants
  * Lithium
  * Selective serotonin and norepinephrine reuptake inhibitors: milnacipran, fluoxetine, paroxetine, nefazodone, citalopram, clovoxamine, escitalopram, flesinoxan, femoxetine, duloxetine, venlafaxine, vilazodone, sibutramine, desvenlafaxine
  * Anticonvulsants: phenytoin, paraldehyde, valproic acid, carbamazepine, trimethadione, phenobarbital, diazepam, chlormethiazole, mephenytoin, ethotoin, paramethadione, phenacemide, mephobarbital, oxcarbazepine, zonisamide, piracetam, vigabatrin, felbamate, gabapentin, beclamide, fosphenytoin, stiripentol, tiagabine, topiramate, pregabalin, lacosamide, rufinamide, caramiphen
  * Antibiotics and antifungals:

    * Fluoroquinolones : such as ofloxacin, norfloxacin, levofloxacin
  * Other agents: teriflunomide, cyclosporine, tacrolimus, ginkgo, gossypol, meadowsweet, feverfew, beta glucan, pentosan, pentoxifylline, cilostazol, erlotinib, pemetrexed, methotrexate, pralatrexate
* Individuals with uncontrolled renal insufficiency or renal failure
* History of allergic reactions attributed to naproxen
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, uncontrolled hypertension, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant, breast-feeding, or women of childbearing potential unwilling to use a reliable contraceptive method; pregnant women are excluded from this study because naproxen/NSAIDs is an agent with the potential for teratogenic or abortifacient effects; because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with naproxen, breastfeeding should be discontinued if the mother is treated with naproxen

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2014-01-27 (Actual); Primary Completion 2019-10-25 (Actual); Study Completion 2021-01-05 (Actual)

PRIMARY OUTCOMES:
Change in PGE2 concentration levels in normal colorectal mucosa | Baseline to 6 months
  Response will be defined as >= 30% reduction in PGE2 levels. Pairwise comparisons by the two-sample t-test among the three groups (low-dose versus control, high-dose versus control, and high-dose versus low-dose) will be used. The calculation adjusts for 3 multiple comparisons using the Bonferroni correction to achieve a two-sided 5% type I error. The point estimate and the 95% exact confidence interval for the response rate will be calculated in each arm.
Minimal biologically effective dose of naproxen that induces a modulation of PGE2 levels | Up to 6 months
Incidence of toxicity | Up to 6 months
  Will be graded according to National Cancer Institute Common Criteria for Adverse Events version 4.0. Descriptive statistics will be used to monitor the type and grade of toxicities. The frequency of toxicities will be compared between the placebo and naproxen groups.

SECONDARY OUTCOMES:
Naproxen concentrations in plasma samples | 6 months
  A t-test or the Wilcoxon rank sum test will be applied for the pairwise comparison of the changes of continuous markers among groups.
Naproxen concentrations in normal colorectal mucosa | 6 months
  A t-test or the Wilcoxon rank sum test will be applied for the pairwise comparison of the changes of continuous markers among groups.
PGE-M levels in urine samples | 6 months
  A t-test or the Wilcoxon rank sum test will be applied for the pairwise comparison of the changes of continuous markers among groups.
Change in number of polyps observed in the rectosigmoid area | Baseline to 6 months
  A t-test or the Wilcoxon rank sum test will be applied for the pairwise comparison of the changes of continuous markers among groups.
Changes in the microRNA profile of the normal colorectal mucosa | Baseline to 6 months
  Bioinformatic methods such as the beta-uniform mixture (BUM) model to account for multiple testing by controlling the false discovery rate (FDR), the Wilcoxon rank-sum test with empirical Bayes, and the significance analysis of microarrays (SAM) with the control of the FDR will be applied using the Object-Oriented Microarray and Proteomic Analysis (OOMPA) program.
Changes in gene expression mRNA profiles of the normal colorectal mucosa | Baseline to 6 months
  Bioinformatic methods such as the BUM model to account for multiple testing by controlling the FDR, the Wilcoxon rank-sum test with empirical Bayes, and the SAM with the control of the FDR will be applied using the OOMPA program.
Changes in the mutational rate of the normal colorectal mucosa | Baseline to 6 months
  Bioinformatic methods such as the BUM model to account for multiple testing by controlling the FDR, the Wilcoxon rank-sum test with empirical Bayes, and the SAM with the control of the FDR will be applied using the OOMPA program.
Changes in the microbiome of the normal colorectal mucosa | Baseline to 6 months
  Bioinformatic methods such as the BUM model to account for multiple testing by controlling the FDR, the Wilcoxon rank-sum test with empirical Bayes, and the SAM with the control of the FDR will be applied using the OOMPA program.
Changes in the PGF2, PGD2, Thromboxane B2, 9a11b-PGF2a and 6-KetoPGF1a levels of the colorectal tissue | Baseline to 6 months
  Bioinformatic methods such as the BUM model to account for multiple testing by controlling the FDR, the Wilcoxon rank-sum test with empirical Bayes, and the SAM with the control of the FDR will be applied using the OOMPA program.
Changes in the stem cell and epithelial differentiation marker levels | Baseline to 6 months
  Bioinformatic methods such as the BUM model to account for multiple testing by controlling the FDR, the Wilcoxon rank-sum test with empirical Bayes, and the SAM with the control of the FDR will be applied using the OOMPA program.
Changes in the number and type of immune and mesenchymal cells recruited to the colorectal mucosa | Baseline to 6 months
  Will be assessed by using a multiplex platform based on imaging cell cytometry (IMC) in a tissue microarray (TMA).

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo Vilar-Sanchez, Principal Investigator — M.D. Anderson Cancer Center
Locations (4):
- United States (4):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - M D Anderson Cancer Center, Houston, Texas
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah

REFERENCES:
- [Derived] Reyes-Uribe L, Wu W, Gelincik O, Bommi PV, Francisco-Cruz A, Solis LM, Lynch PM, Lim R, Stoffel EM, Kanth P, Samadder NJ, Mork ME, Taggart MW, Milne GL, Marnett LJ, Vornik L, Liu DD, Revuelta M, Chang K, You YN, Kopelovich L, Wistuba II, Lee JJ, Sei S, Shoemaker RH, Szabo E, Richmond E, Umar A, Perloff M, Brown PH, Lipkin SM, Vilar E. Naproxen chemoprevention promotes immune activation in Lynch syndrome colorectal mucosa. Gut. 2021 Mar;70(3):555-566. doi: 10.1136/gutjnl-2020-320946. Epub 2020 Jul 8. PMID 32641470